CLINICAL TRIAL: NCT04123535
Title: Focused Ultrasound to Promote Immune Responses for Undifferentiated Pleomorphic Sarcoma
Acronym: HIFU-UPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Bucknor (Other)
Collaborators: Focused Ultrasound Foundation (Other); InSightec-TxSonics (Industry)
Responsible Party: Sponsor-Investigator, Matthew Bucknor, Assistant Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19653; NCI-2019-06737 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Undifferentiated Pleomorphic Sarcoma
Keywords: Focused Ultrasound; Sarcoma
MeSH Terms: conditions — Histiocytoma, Malignant Fibrous; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Undifferentiated Pleomorphic Sarcoma (UPS) (Experimental): All enrolled participants will be scheduled to receive pre-operative MRgFUS with the ExAblate 2000/2100 MRgFUS system 1-4 weeks prior to surgical resection of their tumor or approximately 2 weeks after a pre-procedure biopsy of the metastatic tumor target depending on diagnosis at enrollment. For patients enrolled with metastatic disease, pre and post-MRgFUS biopsy samples will be obtained.
  Interventions: Device: ExAblate 2000/2100 Magnetic Resonance-guided Focused Ultrasound (MRgFUS)

INTERVENTIONS:
Device: ExAblate 2000/2100 Magnetic Resonance-guided Focused Ultrasound (MRgFUS) — The ExAblate 2100 MRgFUS system (InSightec, Inc., Dallas, Texas, USA) is a noninvasive thermal ablation device fully integrated with an MR imaging system and used for the ablation of soft tissue and bone.14-16 The ExAblate combines a focused ultrasound surgery (FUS) delivery system and a conventional diagnostic 3T Magnetic Resonance (MR) scanner. The ExAblate systems provide a real-time therapy planning algorithm, thermal dosimetry, and closed-loop therapy control. The ExAblate transducer device is an integrated component of the MR table
  Other Names: ExAblate 2000/2100; MRgFUS

SUMMARY:
This study is a single site, single-arm, feasibility study to evaluate the safety and efficacy of MRgFUS using the ExAblate 2100 System for the partial ablation of undifferentiated pleomorphic sarcomas.

DETAILED DESCRIPTION:
A total of 20 adult participants will be treated with MRgFUS through this study. A matched comparison group of archived samples from patients with UPS who have not received focused ultrasound will be used as a control group to further evaluate the secondary endpoints (stratified and matched for age, sex, and history of neoadjuvant chemotherapy). All patients enrolled will receive timely standard of care surgical resection, as clinically indicated. For patients enrolled with metastatic disease pre- and post-MRgFUS biopsy samples will be obtained

PRIMARY OBJECTIVE:

I. To evaluate the overall rate and severity of adverse events following MRgFUS of newly diagnosed or metastatic undifferentiated pleomorphic sarcoma.

SECONDARY OBJECTIVES:

I. To measure possible immune response effects related to MRgFUS by serial serological analysis with flow cytometry panels (T-cell, natural killer cell, myeloid panels).

II. To measure possible immune response effects related to MRgFUS by multiplex immunohistochemistry assays of resected tumor specimens (CD3, CD4, CD8, CD19, CD68, FOXP3, PD-1, PD-L1, CD45) as well as RNA sequencing.

III. To compare possible immune response effects in patients receiving MRgFUS prior to either surgical resection or follow-up biopsy of undifferentiated pleomorphic sarcoma to either 1) a comparison group of archived samples from patients who have had resection of UPS but did not have pre-operative focused ultrasound (for patients with newly diagnosed local disease or 2) individual pre-MRgFUS biopsy analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women >= 18 years old.
2. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0-1.
3. Subjects must have either 1) a biopsy-proven new diagnosis of undifferentiated pleomorphic sarcoma (UPS) (within the last 6 months) or 2) a lesion highly suspicious for metastatic UPS based on CT or MRI imaging (within the last 6 months).
4. Target tumor >= 2 cm in maximum diameter and <= 20 cm in maximum diameter.
5. Target tumor accessible to the ExAblate device in the soft tissues of the chest, abdomen, pelvis, or upper or lower extremities.
6. Target tumor must be > 1 cm from any critical structure. Critical structures are defined as skin, major nerve/vascular bundles, nerve roots, any solid organ, and any portion of the bowel.
7. Target tumor must be clearly visible by non-contrast magnetic resonance imaging (MRI)
8. For patients with newly diagnosed, not previously treated UPS, tumor must be deemed to be surgically resectable by tumor board documentation or surgeon's note.
9. To clarify, patient's being treated with institutional standard neoadjuvant chemotherapy may be included in this study if all other inclusion/exclusion criteria are met.

   * Note: There has never been a prospective study comparing patients receiving chemotherapy to those not receiving chemotherapy in the neoadjuvant setting for soft tissue sarcoma. Our local institutional standard is to treat patients with neoadjuvant chemotherapy prior to surgical resection when tumors are > 5 cm in maximal dimension and within deep muscular compartments. Our institutional standard is to treat patients with doxorubicin plus ifosfamide for younger patients (typically <50 years old) and gemcitabine plus taxotere for older patients (typically >= 50 years old).

Exclusion Criteria:

1. Subjects requiring systemic treatment with corticosteroids or other immunosuppressive medications within 14 days of Magnetic Resonance-guided Focused Ultrasound (MRgFUS) treatment date.
2. History of interstitial lung disease or other active malignancy (may confound immune response results).
3. History of previous malignancies (except non-melanoma skin cancers) (may confound immune response results).
4. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to grade 1 (NCI CTCAE version 4) or baseline.
5. Subjects must have recovered from the effects of major surgery or significant trauma at least 14 days before the study procedure.
6. Subjects with an acute medical condition expected to hinder them from completing the study, unstable cardiovascular status, and severe cerebrovascular disease.
7. Treatment with any investigational agent within 28 days of the treatment procedure.
8. Any absolute contraindications for study magnetic resonance imaging (MRI) per standard University of California, San Francisco (UCSF) departmental MRI safety guidance (https://radiology.ucsf.edu/patient-care/patient-safety/mri) and additionally:

   * Metal in other parts of body that will cause safety issues
   * Claustrophobia
   * Weight > 400 pounds (lb) or 181.4 kilograms (kg).
   * Pregnancy
   * Known intolerance or allergy to magnetic resonance (MR) contrast agent (gadolinium chelates)
9. Unable to safely receive anesthesia/sedation for the treatment, or known intolerance or allergy to medications used for sedation/anesthesia.
10. Unable to verbally communicate with the investigator and staff.
11. For Group 1 Patients (newly diagnosed disease) only: Have received neoadjuvant radiotherapy or planning to receive neoadjuvant radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with reported Device-Related Adverse Events | Approximately 1-4 months
  Proportion of participants with device-related adverse events will be determined by evaluating the incidence and severity of any device-related complications from the treatment day visit through the time of surgery or last post-treatment point. Patients will be followed for any reported adverse events following MRgFUS, per the Common Terminology Criteria for Adverse Events version 5.0

SECONDARY OUTCOMES:
Percent change between baseline and post-treatment T-cell populations | Approximately 1-4 months
  Blood samples obtained at 1 week prior to MRgFUS and at 1 week post MRgFUS will be sent to the University of California, San Francisco (UCSF) Cancer Immunotherapy Lab. Flow cytometry panels will be performed to evaluate T-cell populations. Percent change between baseline and post-treatment samples will be calculated and displayed as a table
Percent change between baseline and post-treatment natural killer cell populations | Approximately 1-4 months
  Blood samples obtained at 1 week prior to MRgFUS and at 1 week post MRgFUS will be sent to the University of California, San Francisco (UCSF) Cancer Immunotherapy Lab. Flow cytometry panels will be performed to evaluate natural killer cell populations. Percent change between baseline and post-treatment samples will be calculated and displayed as a table
Percent change between baseline and post-treatment myeloid cell populations | Approximately 1-4 months
  Blood samples obtained at 1 week prior to MRgFUS and at 1 week post MRgFUS will be sent to the University of California, San Francisco (UCSF) Cancer Immunotherapy Lab. Flow cytometry panels will be performed to evaluate myeloid cell populations. Percent change between baseline and post-treatment samples will be calculated and displayed as a table
Percent change between baseline and post-treatment Cytokine Concentrations | Approximately 1-4 months
  Blood samples obtained at 1 week prior to MRgFUS and at 1 week post MRgFUS. Cytokine concentrations will also be measured. Percent change between baseline and post-treatment samples will be calculated
Presence of Immune Cell Populations in Sarcoma Tissue | Approximately 1-4 months
  The detectable presence of various immune populations in tumor specimens, including populations of CD3, CD4, CD8, CD19, CD68, FOXP3, PD-1, PD-L1, and CD45 positive cells will be determined. RNA sequencing will also be performed.
Immunohistochemistry analyses | Approximately 1-4 months
  Immunohistochemistry analyses in patients with newly diagnosed local UPS will be compared to an archived matched group of patients (matched for age, sex, and history of neoadjuvant chemotherapy) who had resection of UPS without pre-operative MRgFUS. Nanostring digital spatial profiling may also be used for tissue analysis

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bucknor, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No